CLINICAL TRIAL: NCT07044687
Title: A Phase 4 Study of Venetoclax in Combination With Azacitidine in Indian Subjects With Newly Diagnosed Acute Myeloid Leukemia Who Are Ineligible for Standard Induction Therapy
Brief Title: Study to Assess Adverse Events and Change in Disease Activity of Oral Venetoclax in Combination With Subcutaneous (SC) or Intravenous (IV) Azacitidine in Newly Diagnosed Adult Participants With Acute Myeloid Leukemia (AML) Who Are Ineligible for Standard Induction Therapy in India
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M23-826
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML; Venetoclax; Venclexta; Azacitidine; Treatment Naïve AML; Untreated AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax in Combination with Azacitidine (Experimental): Participants will receive venetoclax once daily in increasing doses until the study dose is achieved. Then ventoclaxwill continue once daily thereafter. Participants will receive azacitidine on Day 1-7 of each cycle. The total study duration is approximately 29 months.
  Interventions: Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Venetoclax — Oral Tablet
Drug: Azacitidine — Subcutaneous (SC) Injection
Drug: Azacitidine — Intravenous (IV) Injection

SUMMARY:
Acute myeloid leukemia (AML) is one of the most aggressive blood cancers, with a very low survival rate and few options for participants who are unable to undergo standard induction therapy, the current standard of care. This study will assess the change in disease activity and adverse events in adult participants with acute myeloid leukemia (AML) being treated with of the combination of azacitidine and venetoclax, in India.

The combination of azacitidine and venetoclax is being evaluated in the treatment of acute myeloid leukemia (AML). Participants will receive azacitidine with increasing doses of venetoclax. Around 40 adult participants with a diagnosis of AML will be enrolled in the study at approximately 15 sites in India.

Participants will receive venetoclax oral tablets once daily in increasing doses until the study dose is achieved. Then ventoclax oral tablets will continue once daily thereafter. Azacitidine will be given by subcutaneous (SC) or intravenous (IV) injection on Days 1-7 of each cycle. The total study duration is approximately 29 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of acute myeloid leukemia (AML) diagnosis by 2016 World Health Organization (WHO) criteria, previously untreated, and ineligible for treatment with intensive chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of:

  * 0 to 2 for subject ≥ 75 years of age.
  * 0 to 3 for subject ≥ 18 to 74 years of age.

Exclusion Criteria:

* History of any malignancy within 2 years prior to study entry with exception to those noted in the protocol.
* Have received any investigational drug 30 days prior to the first dose of study drug and have received strong CYP3A inducers within 7 days prior to the initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Treatment Emergent Adverse Events (TEAE)s | Up to Approximately 29 Months
  TEAEs defined as any adverse event (AE) with the onset after the first dose of study drug until 30 days after the last dose of the study drug.
Percentage of Participants with Post-Baseline Laboratory Abnormalities | Up to Approximately 29 Months
  Laboratory abnormalities are defined based on the shifts from baseline to postbaseline laboratory values will be summarized using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Composite Complete Remission (CRc) | Up to Approximately 29 Months
  (CRc) is defined as Complete remission (CR) or complete remission with incomplete marrow recovery (CRi) per the modified International Working Group (IWG) response criteria for AML in participants who received venetoclax and azacitidine combination study treatment.
Composite Complete Remission (CRc) by initiation of Cycle 2 | Up to Approximately 1 Month
  (CRc) is defined as Complete remission (CR) or complete remission with incomplete marrow recovery (CRi) per the modified International Working Group (IWG) response criteria for AML in participants who received venetoclax and azacitidine combination study treatment.
Complete Remission | Up to Approximately 29 Months
  CR is defined as the modified IWG response criteria for AML in participants who received venetoclax and azacitidine combination study treatment.
Overall Survival (OS) | Up to Approximately 29 Months
  OS is defined as the time measured from randomization until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (11):
- India (11):
  - Fortis Memorial Research Institute /ID# 268697, Gurgaon, Haryana
  - Mazumdar Shaw Medical Center /ID# 270677, Bengaluru, Karnataka
  - Regional Cancer Centre /ID# 268785, Thiruvananthapuram, Kerala
  - LMMF's Deenanath Mangeshkar Hospital & Research Center /ID# 268781, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital /ID# 272074, Pune, Maharashtra
  - All India Institute Of Medical Sciences - New Delhi /ID# 268357, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Institute And Research Centre /ID# 268293, New Delhi, National Capital Territory of Delhi
  - All India Institute Of Medical Sciences - Bhubaneswar /ID# 274879, Bhubaneswar, Odisha
  - Apollo Cancer Centre /ID# 268780, Chennai, Tamil Nadu
  - Cancer Institute (Wia) /ID# 268695, Chennai, Tamil Nadu
  - Basavatarakam Indo American Cancer Hospital & Research Institute /ID# 268692, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-826